CLINICAL TRIAL: NCT03633890
Title: A Randomized, Double-Blind, Placebo-Controlled Trial for DaZhu Rhodiola Rosea Capsule in the Treatment of Coronary Artery Disease With Angina Pectoris
Brief Title: DaZhu Rhodiola Rosea Capsule for Coronary Artery Disease With Angina Pectoris
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Anzhen Hospital (Other)
Collaborators: Jiangsu Kangyuan Pharmaceutical Co. Ltd (Unknown)
Responsible Party: Principal Investigator, Shao-Ping Nie, Professor of Medicine, Director, Emergency & Critical Care Center, Beijing Anzhen Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017032
Record Dates: First submitted 2018-08-07; First posted 2018-08-16 (Actual); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DaZhu Rhodiola Rosea Capsule (Experimental)
  Interventions: Drug: DaZhu Rhodiola Rosea Capsule
- DaZhu Rhodiola Rosea Simulation Capsule (Placebo Comparator)
  Interventions: Drug: DaZhu Rhodiola Rosea Simulation Capsule

INTERVENTIONS:
Drug: DaZhu Rhodiola Rosea Capsule — Oral administration, 4 capsules, 3 times a day, for 8 weeks
  Arms: DaZhu Rhodiola Rosea Capsule
Drug: DaZhu Rhodiola Rosea Simulation Capsule — Oral administration, 4 capsules, 3 times a day, for 8 weeks
  Arms: DaZhu Rhodiola Rosea Simulation Capsule

SUMMARY:
This study aims to evaluate the efficacy and safety of traditional Chinese medicine DaZhu Rhodiola Rosea Capsule for treatment of coronary artery disease by observing angina symptoms, exercise capacity, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 75 years old
* Coronary heart disease with grade Ⅱ or Ⅲ stable or unstable angina (≥ 2 times per week), or residual angina-like symptoms 1 month to 1 year post percutaneous coronary intervention (PCI) or 3 months to 1 year post coronary artery bypass surgery (CABG)
* Written informed consent

Exclusion Criteria:

* Acute myocardial infarction within 1 month before admission
* Patients who plan to undergo revascularization in the next 3 months
* Congestive heart failure, acute myocarditis or pericarditis, thrombophlebitis, pulmonary embolism, or severe neurosis within 3 months prior to admission
* Patients with uncontrolled high blood pressure (systolic blood pressure greater than 160 mmHg or diastolic blood pressure greater than 100 mmHg), severe cardiopulmonary insufficiency (cardiac function grade Ⅲ, Ⅳ or left ventricular ejection fraction (LVEF) < 40%), severe arrhythmia (rapid atrial fibrillation and flutter, paroxysmal ventricular tachycardia, degree Ⅱ type Ⅱ and degree Ⅲ atrioventricular block, etc.)
* Severe liver, kidney and hematopoietic system dysfunction or psychosis (serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2 times the normal upper limit, or serum creatinine > 1.5 times the normal upper limit)
* History of bleeding or treatment with warfarin
* Implanted pacemakers
* Pregnant or lactating women
* Allergic to study drugs
* Legal disability (blindness, deafness, dumbness, intellectual disability, mental disability, physical disability)
* Patients who participated in other clinical trials within 3 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2018-08 (Estimated); Primary Completion 2019-02 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Seattle Angina Questionnaire (SAQ) angina frequency | week 8
  Scored from 0 to 100, with higher scores indicating better health status

SECONDARY OUTCOMES:
SAQ angina stability | week 8
  Scored from 0 to 100, with higher scores indicating better health status
SAQ physical limitation | week 8
  Scored from 0 to 100, with higher scores indicating better health status
SAQ treatment satisfaction | week 8
  Scored from 0 to 100, with higher scores indicating better health status
SAQ disease perception | week 8
  Scored from 0 to 100, with higher scores indicating better health status
Walking distance by 6-minute walking test | week 8
Frequency of angina | week 8
visual analogue scale (VAS) score | week 8
  Scored from 0 to 10, with higher scores indicating worse health status
36-item Short Form Health Survey (SF-36) score | week 8
  Scored from 36 to 180, with higher scores indicating better health status

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Anzhen Hospital, Capital Medical University, Beijing, China